CLINICAL TRIAL: NCT00018837
Title: Brief Hospitalization for Schizophrenia: Strategies to Improve Treatment Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Organization: VA Office of Research and Development (U.S. Federal Agency)
Model: Parallel
Other Study IDs: MHBS-010-98S
Record Dates: First submitted 2001-07-03; First posted 2001-07-05 (Estimated); Last update posted 2009-01-21 (Estimated); Status verified 2004-12

CONDITIONS: Schizophrenia; Schizophrenic Disorder
MeSH Terms: conditions — Schizophrenia

INTERVENTIONS:
Behavioral: Community Re-Entry Program: What is Schizophrenia

SUMMARY:
The goal of this research program is to implement a series of psychoeducational training classes designed to teach individuals with schizophrenia the importance of medication treatment, how to identify and manage medication side effects, and how to make appointments and emergency plans. The skills taught to the research subjects will lead to demonstrable increases (compared to the control group) in adherence to both the prescribed medication regimen and scheduled outpatient appointments and thereby cause a decrease (again compared to the control group) in rehospitalization rates and bed-days during subsequent twelve months following the intervention. A secondary objective of this work is that if the CREP program is successful and/or illness education is effective, the data will be able to disseminated throughout the VISN 22 via the recently awarded Mental Illness Research Education and Clinical Center (MIRECC) program.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years of age.
2. DSM IV diagnosis of schizophrenia or schizoaffective disorder.
3. Competent to give informed consent.
4. Previously participated in "Brief Hospitalization for Schizophrenia: Strategies to Improve Treatment Outcome" Principal Investigator. Donna Wirshing, M.D.

Exclusion Criteria:

1. Physical or cognitive impairment of such severity as to adversely affect the validity of clinical ratings or impair capacity to give informed consent.
2. History of substantial substance dependence 6 months prior to the study.
3. Patients at high risk of suicide or other directed violence.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-04; Study Completion 2001-03

CONTACTS AND LOCATIONS:
Locations (1):
- VA Greater Los Angeles Healthcare System, Los Angeles, California, United States